CLINICAL TRIAL: NCT06542367
Title: Trans Canal Tympanoplasty With Local Anesthesia Using Fat Graft and "TachoSil"
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Yoni Evgeni Gutkovich, Doctor, HaEmek Medical Center, Israel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0047-24-EMC
Record Dates: First submitted 2024-08-01; First posted 2024-08-07 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Tympanic Membrane Perforation
Keywords: Tympanoplasty
MeSH Terms: conditions — Tympanic Membrane Perforation | interventions — TachoSil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Transcanal tympanoplasty under local anasthesia with fat graft and "Tachosil" (Experimental): eligibale participatns with chronic tympanic membrane perforation will be offered to participate.
  Under local anesthesia, subcutaneous fat from the neck will be harvested. After that trimming of the perforation edges, planting the fat graft medial to the tympanic membrane and placement of the "Tachosil" on top of the fat graft.
  gelfoam is placed lateral to the tympanic membrane fo fill the ear canal. follow-up will be held at 2, 4-6 and 12 month following the procedure, with audiometric and otological evaluation
  Interventions: Procedure: Tympanoplasty performed under local anesthesia using fat graft and "Tachosil".

INTERVENTIONS:
Procedure: Tympanoplasty performed under local anesthesia using fat graft and "Tachosil". — Under local anesthesia, subcutaneous fat from the neck will be harvested. After that trimming of the perforation edges, planting the fat graft medial to the tympanic membrane and placement of the "Tachosil" on top of the fat graft.
  gelfoam is placed lateral to the tympanic membrane to fill the ear canal. follow-up will be held at 2, 4-6 and 12 months following the procedure, with audiometric and otological evaluation

SUMMARY:
Eligible participants with chronic tympanic membrane perforation (>6 month) will be given a detailed description and offered to participate in the study.

the study investigates the efficacy of trans canal tympanoplasty with local anesthesia using fat pad and "Tachosil". Participants will be followed for 1 year after the procedure with otological examination and successive hearing evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Chronic tympanic membrane perforation (>6 months).
* Central tympanic membrane perforation.
* Air bone gar of 35 dB or lower at the operated ear.
* No active otorrhea in the operated ear in the preceding 3 month prior to the procedure.
* No evidence of a retraction pocket and no suspicion for a cholesteatoma.

Exclusion Criteria:

* Known ossicular chain dysfunction
* The tympanic membrane perforation edges are not accessible/visualized transcanal
* Pregnancy
* Allergy to lidocaine

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
closure of tympanic membrane perforation | 1 year following the procedure
  the effectiveness of the tympanoplasty using far graft and "Tachosil" will be evaluated - whether close of tympanic membrane perforation occured.

SECONDARY OUTCOMES:
Hearing results following tympanoplasty - Speech recognition threshold | 1 year following the procedure
  SRT (Speech recognition threshold) in dB (Decibel) will be evaluated pre and post tympanoplasty using an audiogram.
Hearing results following tympanoplasty - Pure Tone Average | 1 year following the procedure
  PTA air and PTA bone (Pure Tone Average) in dB (Decibel) will be evaluated pre and post tympanoplasty using an audiogram.
Hearing results following tympanoplasty - air bone gap. | 1 year following the procedure
  Air-bone gap in dB (Decibel) will be evaluated pre and post tympanoplasty using an audiogram.

IPD SHARING:
Plan to Share IPD: Undecided